CLINICAL TRIAL: NCT04622202
Title: The Effects Of Pre-emptive Single Oral Dose Pregabalin on Attenuating Maternal Anxiety And Stress Response To Intubation During Caesarean Section
Brief Title: Pre-emptive Pregabalin on Attenuating Maternal Anxiety And Stress Response To Intubation During Caesarean Section
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sara mohamed Abdelnaby, lecturer of anaesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6408
Record Dates: First submitted 2020-10-27; First posted 2020-11-09 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Anxiety State; Sedation
MeSH Terms: conditions — Anxiety Disorders | interventions — Pregabalin; Geritol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pregabalin (Active Comparator): oral capsule pregabalin 150 mg.
  Interventions: Drug: Pregabalin 150mg
- multivitamin (Placebo Comparator): oral multivitamin capsule.
  Interventions: Drug: multivitamin

INTERVENTIONS:
Drug: Pregabalin 150mg — oral capsule pregabalin 150 mg.
  Other Names: Lyrica
  Arms: pregabalin
Drug: multivitamin — oral placebo in the form of oral multivitamin capsule.
  Other Names: Placebo
  Arms: multivitamin

SUMMARY:
There is exaggerated neuroendocrine stress response to laryngoscopy and endotracheal intubation during the Induction to anesthesia-delivery (I-D) period under light anesthesia. Mechanical stimulation of laryngeal proprioceptors elicits increased secretion of cortisol and catecholamine with subsequent elevation of blood pressure from 40 to 50 % and heart rate up to 20 % during direct laryngoscopy and endotracheal intubation

DETAILED DESCRIPTION:
The sample size was calculated using OPEN EPI program assuming that the mean visual analogue scale anxiety score was 49.3±14.1 among oral pregabalin group and was 58.6± 14.4 among Placebo group (8) so at power of study 80% confidence interval 95%, the sample size was calculated to be 74 cases (37in each group

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-38 years old.
* Pregnant Female with a singleton fetus of at least 36 weeks of gestation.
* American Society of Anesthesiologist Physical status: 1& II.
* Body Mass Index (BMI) (25-30kg/m²).
* Type of operations: elective caesarean section under general anesthesia.
* Written informed consent from the parturient.

Exclusion Criteria:

* Altered mental state.
* Women with known history of allergy to pregabalin.
* Women with uncontrolled diabetes mellitus, bleeding, coagulation disorders, Hepatic, renal, Cardiovascular, respiratory disease and neuropsychiatric disorders.
* Patients receiving anticonvulsants, antidepressants.
* Pregnancy induced hypertension, intrauterine growth restriction or fetal compromise

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
preoperative maternal anxiety changes | change from baseline at 60 minutes after giving drug preoperative.
  Anxiety by State-Trait Anxiety Inventory (STAI) questionnaire before drug administration and 60 minutes after giving drug (pre-induction).

SECONDARY OUTCOMES:
Number of participant with changes in level of consciousness | at 60 minutes preoperative
  changes in level of consciousness of participant by Alert, verbal response, pain response and unresponsive (AVPU) scale 60 minutes after giving drug (pre-induction).
  Alert: The patient is aware of the examiner and can respond to the environment around them on their own. The patient can also follow commands, open their eyes spontaneously, and track objects.
  Verbally Responsive: The patient's eyes do not open spontaneously. The patient's eyes open only in response to a verbal stimulus directed toward them. The patient is able to react to that verbal stimulus directly and in a meaningful way.
  Painfully Responsive: The patient's eyes do not open spontaneously. The patient will only respond to the application of painful stimuli by an examiner. The patient may move, moan, or cry out directly in response to the painful stimuli.
  Unresponsive: The patient does not respond spontaneously. The patient does not respond to verbal or painful stimuli.
Heart rate | at baseline, 0 (at intubation) 1, 3, 5, 10 and 15 minutes after intubation.
  Heart rate will be recorded preoperative baseline, 0 (at intubation) 1, 3, 5, 10 and 15 minutes after intubation.
mean arterial blood pressure | at baseline, 0 (at intubation) 1, 3, 5, 10 and 15 minutes after intubation.
  mean arterial blood pressure
Serum glucose | preoperative and at 10 minutes after intubation.
  Serum glucose level will be recorded preoperative and at 10 minutes after intubation.
cortisol level | preoperative and at 10 minutes after intubation.
  cortisol level will be recorded preoperative and at 10 minutes after intubation.
Baby Apgar score | at 1 and 5 minutes after delivery
  Apgar score at 1 and 5 min after delivery Apgar Scoring
  Apgar Sign 2 1 0 Appearance (skin color) Normal color all over (hands and feet are pink) Normal color (but hands and feet are bluish) Bluish-gray or pale all over Pulse (heart rate) Normal (above 100 beats per minute) Below 100 beats per minute Absent (no pulse) Grimace ("reflex irritability") Pulls away, sneezes, coughs, or cries with stimulation Facial movement only (grimace) with stimulation Absent (no response to stimulation) Activity (muscle tone) Active, spontaneous movement Arms and legs flexed with little movement No movement, "floppy" tone Respiration (breathing rate and effort) Normal rate and effort, good cry Slow or irregular breathing, weak cry Absent (no breathing)
  A baby who scores a 7 or above on the test is considered in good health.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Abdel Naby, M.D, Principal Investigator — Zagazig University
Locations (1):
- Sara Mohamed Abdel Nabi, Zagazig, Egypt